CLINICAL TRIAL: NCT00584935
Title: Phase I/II Clinical Trial Evaluating Rituximab in Ocular Cicatricial Pemphigoid
Brief Title: Clinical Trial Evaluating Rituximab in Ocular Cicatricial Pemphigoid
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry); Biogen (Industry)
Responsible Party: Principal Investigator, Craig Elmets, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F060213003
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Ocular Cicatricial Pemphigoid
Keywords: Pemphigoid; Blistering Diseases; Blindness; Autoimmune; Rituximab
MeSH Terms: conditions — Pemphigoid, Benign Mucous Membrane; Pemphigoid, Bullous; Blindness | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab (Experimental): The Rituximab dose is 1000 mg (1gm) given as an IV infusion every two weeks for 2 doses (Days 1 and 15).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — The Rituximab dose is 1000mg (1gm) given as an IV infusion every two weeks for 2 doses (days 1 and 15).

SUMMARY:
Cicatricial pemphigoid is an autoimmune blistering disease which affects the skin, mucous membranes, and, in a small subset of patients, the eye. Progressive ocular disease can lead to irreversible damage and blindness. Conventional treatments include systemic steroids, dapsone, and immunosuppressive agents. These treatments, however, are not successful with all patients. Rituximab has been very effective in the treatment of other autoimmune disorders, and has recently been shown to be effective for autoimmune blistering pemphigus. We propose that it will also be effective in the treatment of cicatricial pemphigoid.

DETAILED DESCRIPTION:
Cicatricial pemphigoid is an autoimmune blistering disease which can affect the skin, mucous membranes, and, in a small subset of patients, the eyes. Progressive ocular disease can lead to irreversible damage and blindness. Conventional treatments have included high dose systemic steroids, dapsone, and immunosuppressive agents such as azathioprine, methotrexate, cyclophosphamide, and mycophenolate mofetil. However, there are a subgroup of patients who fail to respond to these treatments, develop intolerable side effects, or have contraindications to their use. Patients may also develop resistance to these conventional treatment modalities. For these reasons, alternative treatment modalities are needed. Rituximab has been very effective in the treatment of other autoimmune disorders. It has recently been shown to be effective in the treatment of another autoimmune blistering disorder known as pemphigus. We thus propose that Rituximab will be effective in the treatment of cicatricial pemphigoid.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ocular cicatricial pemphigoid (symptoms of conjunctivitis, irritation, burning, increased lacrimation, photophobia, dryness of the eyes along with conjunctival inflammation, trichiasis, and scarring
2. One of the following:

   * Failed response to the use of one or more conventional treatments for a minimum of 10 weeks; or
   * Minimal conventional medication doses, with a significant adverse effects, contradiction to use, or progressive disease despite treatment
3. Adults age 19 and older
4. Adequate renal function as indicated by serum creatinine levels less than 1.5

Exclusion Criteria:

1. known hypersensitivity to rituximab or its components
2. Age less than 19 years
3. Any other condition deemed by the investigator to be a significant hazard to the subject if the investigational therapy were initiated.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Elmets, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three patients were recruited from the investigator's practice.
Pre-assignment Details: Subjects must meet inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Rituximab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Evidence of Further Scarring (Fosters Staging) at 16 Weeks
Description: Stages Characteristics I Subconjunctival scarring and fibrosis II Fornix foreshortening (a-d describes % loss of inferior fornix depth)
  1. 0-25%
  2. 25-50%
  3. 50-75%
  4. 75-100% III Presence of symblepharon and number (n) (a-d describes % of horizontal involvement by symblepharons and n is the number of symblepharons countable)
  a. 0-25% b. 25-50% c. 50-75% d. 75-100% IV Ankyloblepharon, frozen globe
Time Frame: 16 weeks
Population: The data for this Outcome was not collected and due to the length of time, the records have been destroyed.
Arm/Group | Rituximab
Number analyzed (Participants) | 0

2. Primary Outcome: 2. The Proportion of Patients That Experience a Grade 3, Grade 4, or Grade 5 Toxicity Based Reaction on the NCI-CTC System at the Time of Their Infusions and During Follow-up Visits.
Time Frame: 16 weeks
Population: The data for this Outcome was not collected and due to the length of time, the records have been destroyed.
Arm/Group | Rituximab
Number analyzed (Participants) | 0

3. Secondary Outcome: 1. Stability of Visual Acuity (Snellen's Test) at 16 Weeks
Time Frame: 16 weeks
Population: The data for this Outcome was not collected and due to the length of time, the records have been destroyed.
Arm/Group | Rituximab
Number analyzed (Participants) | 0

4. Secondary Outcome: 2. Stability of Visual Acuity (Snellen's Test) at 24 Weeks
Time Frame: 24 weeks
Population: The data for this Outcome was not collected and due to the length of time, the records have been destroyed.
Arm/Group | Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Genentech closed trial before site was able to enroll 5 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator is required to submit the final manuscript to the sponsor prior to publication. The sponsor may suggest changes but investigator retains editorial rights.